CLINICAL TRIAL: NCT04780451
Title: 12 Weeks of Omega-3 Supplementation Combined With Endurance Training Improve Running Economy in Recreational Runners. The Potential Role of the Myokines-NO Pathway.
Brief Title: Omega-3 Supplementation Combined With Endurance Training Improve Running Economy in Recreational Runners.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018/31/N/NZ7/02962
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Effect of Omega-3 Supplementation on Exercise Performance and Muscle Tissue Functions
Keywords: omega-3; supplementation; endurance training; running

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega (Experimental)
  Interventions: Dietary Supplement: Omega-3 supplementation in recreational runners
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Omega-3 supplementation in recreational runners

INTERVENTIONS:
Dietary Supplement: Omega-3 supplementation in recreational runners — Male recreational runners participated in 12 weeks of endurance training combined with omega-3 fatty acids supplementation. Before starting and at the end of the 12-week cycle, the runners performed an increasing intensity treadmill test where oxygen uptake and VO2 peak were assessed.

SUMMARY:
Recreational male runners participated in 12 weeks training and omega-3 supplementation programme. Before starting and at the end of the 12-week cycle, the runners performed an increasing intensity treadmill test where oxygen uptake and VO2 peak were assessed.

DETAILED DESCRIPTION:
40 healthy, recreational male runners participated in 12 weeks training and supplementation programme. The training protocol was built based on undulatory load manipulation 3:1, which was suggested to be effective to prevent overtraining and stress due to oscillations between volume/intensity. Throughout the study all participants took 4 identical-looking capsules per day (2 in the morning and 2 in the evening) containing either omega-3 fatty acids or medium chain triglycerides as placebo in total amount of 4g of fat per day. Before starting and at the end of the 12-week cycle, the runners performed an increasing intensity treadmill test where oxygen uptake and VO2 peak were assessed. Additionally, blood was collected to determine the concentrations of selected proteins (including eNOS, irisin, adiponectin) that may be associated with potential changes in participants' oxygen uptake during the treadmill test.

ELIGIBILITY:
Inclusion Criteria:

* non smoking
* no chronic diseases
* no supplements and medicines
* personal best in 10km run between 35 and 59 min at the turn of 2016 and 2020 y

Exclusion Criteria:

-

Ages: 29 Years to 42 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
changes in oxygen consumption during running test | between 10 and 25 minutes of the running test

CONTACTS AND LOCATIONS:
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland